CLINICAL TRIAL: NCT04203758
Title: High Fiber Rye Foods for Body Weight and Body Fat Reduction - The RyeWeight2 Study, a Randomized Controlled Trial.
Brief Title: High Fiber Rye Foods for Body Weight and Body Fat Reduction
Acronym: RyeWeight2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Responsible Party: Principal Investigator, Rikard Landberg, Professor, Chalmers University of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RW2
Record Dates: First submitted 2019-12-13; First posted 2019-12-18 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wholegrain rye products with a high content of dietary fiber (Experimental): Cereal products based on wholegrain rye
  Interventions: Other: Cereal products based on rye
- Refined wheat products with a low content of dietary fiber (Active Comparator): Cereal products based on refined wheat
  Interventions: Other: Cereal products based on wheat

INTERVENTIONS:
Other: Cereal products based on rye — Participants will receive a fixed amount of rye based cereals products, corresponding to approx 650 kcal/day.
  Arms: Wholegrain rye products with a high content of dietary fiber
Other: Cereal products based on wheat — Participants will receive a fixed amount of wheat based cereals products, corresponding to approx 650 kcal/day.
  Arms: Refined wheat products with a low content of dietary fiber

SUMMARY:
The overall aim of this study is to investigate whether a diet rich in rye fiber from wholegrain rye, compared to refined wheat, as part of a hypo-caloric diet leads to larger weight loss and lower body fat content after 12 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 30-70 y
* BMI 27-35 kg/m2
* Hemoglobin ≥117g/l for women and for men ≥134g/l
* Thyroid stimulating hormone (TSH) ≤4.30 mIU/L
* Low density lipoprotein (LDL) cholesterol ≤5.30 mmol/L
* Triglycerides ≤2.60 mmol/L
* Signed informed consent

Exclusion Criteria:

* Blood donation or participation in a clinical study with blood sampling within 30 days prior to screening visit and throughout the study
* Unable to satisfactorily complete the 3-day weighted food record between screening visits.
* Unable to lose ≥0.5 kg during the run-in period for men and women not having menstruation during the run-in period
* Increased body weight, despite reported adherence to dietary intake for women with menstruation during the run-in period.
* Using nicotine products on a daily basis (incl. chewing gum, patches, snus etc.)
* Using e-cigarettes (regardless of nicotine content)
* Following any weight reduction program or having followed one during the last 6 months prior to visit 1.
* Diastolic blood pressure 105 mmHg or more at visit 1
* Systolic blood pressure 160 mmHg or more at visit 1
* History of stomach or gastrointestinal conditions (Inflammatory bowel disease, Crohn's disease, malabsorption, colostomy, bowel resection, gastric bypass surgery etc.)
* More than 10 hours physical activity per week
* History of heart failure or heart attack within 1 year prior to screening
* Having type I diabetes
* Receiving pharmacological treatment for type II diabetes (treatments based on life style interventions are acceptable, as long as they are compatible with the study protocol)
* Previous gastrointestinal surgery, with the exception of minor surgeries such removal of appendix or gall bladder at least 6 months prior to screening.
* Thyroid disorder
* History of eating disorder
* History of drug or alcohol abuse
* Stroke or transient ischemic attack (TIA) within 1 year prior to screening
* Consumption of drugs aimed at weight management or drugs affecting body weight to a degree that is considered unsuitable for study participation by responsible physician.
* Pregnant, lactation or planning a pregnancy within the timeframe of the study. Pregnancy must have ended at least 6 months prior to screening, and lactation must have ended at least 1 month prior to screening.
* Food allergies or intolerances preventing consumption of any products included in the study
* Strict vegetarian (participants must be able to consume the standardized meals used for appetite assessment)
* Unable to sufficiently understand written and spoken Swedish to provide written consent and understand information and instructions from the study personal.
* Lack of suitability for participation in the study, for any reason, as judged by the medical doctor or PI.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Investigate if there is a difference in body weight at week 12 | 12 weeks
  Measured on a scale
Investigate if there is a difference in body fat mass at week 12 | 12 weeks
  Measured by dual energy x-ray absorptiometry

SECONDARY OUTCOMES:
Investigate if there are differences in subjective appetite ratings | 0 weeks, 6 weeks and 12 weeks.
  Measured by visual analogue scale (assessing hunger fullness and desire to eat), throughout a whole day (8:00-21:00), at baseline, week 6 and week 12.
Investigate if differences in primary endpoints (body weight) are apparent at week 6 | 6 weeks
  Measured on a scale
Investigate if differences in primary endpoints (fat mass) are apparent at week 6 | 6 weeks
  Measured by dual energy x-ray absorptiometry
Investigate if lean body mass differs between intervention groups after 6 and 12 weeks of intervention | 6 weeks and 12 weeks
  Measured by dual energy x-ray absorptiometry
Investigate if abdominal fat mass differs between intervention groups after 6 and 12 weeks of intervention | 6 weeks and 12 weeks
  Measured by dual energy x-ray absorptiometry
Investigate if fasting plasma triglycerides differ between groups | 6 weeks and 12 weeks
Investigate if fasting plasma low-density lipoprotein cholesterol differ between groups | 6 weeks and 12 weeks
Investigate if fasting plasma high-density lipoprotein cholesterol differ between groups | 6 weeks and 12 weeks
Investigate if fasting plasma total cholesterol differ between groups | 6 weeks and 12 weeks
Investigate if fasting plasma glucose differ between groups | 6 weeks and 12 weeks
Investigate if fasting serum insulin differ between groups | 6 weeks and 12 weeks
Investigate if C-reactive protein differ between groups | 6 weeks and 12 weeks
Investigate if gut microbiota composition is affected by the intervention | 6 weeks and 12 weeks
  Gut microbiota composition will be analyzed using 16S ribosomal ribonucleic acid (rRNA) sequencing
Investigate if hip circumference differ between intervention groups | 6 weeks and 12 weeks
Investigate if waist circumference differ between intervention | 6 weeks and 12 weeks
Investigate if sagittal height differ between intervention groups | 6 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Landberg, PhD, Principal Investigator — Chalmers University of Technology
Locations (1):
- Chalmers University of Technology, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No